CLINICAL TRIAL: NCT05202002
Title: Decreasing the Incidence of Post-partum Type II Diabetes Mellitus in Gestational Diabetes Population- Prospective Randomized Controlled Trial
Brief Title: Decrease Type II Diabetes in Gestational Diabetes Population
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Carmel Medical Center (Other)
Responsible Party: Principal Investigator, Nadav Cohen, Principal Investigator, Carmel Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: CMC-20-0041-CTIL
Record Dates: First submitted 2022-01-08; First posted 2022-01-21 (Actual); Last update posted 2022-02-04 (Actual); Status verified 2022-01

CONDITIONS: Gestational Diabetes; Diabetes Mellitus, Type 2; Breastfeeding; Diabetes Mellitus, Type 1; Impaired Glucose Tolerance
MeSH Terms: conditions — Diabetes, Gestational; Diabetes Mellitus, Type 2; Breast Feeding; Diabetes Mellitus, Type 1; Glucose Intolerance | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Educational video (Active Comparator): Participants will receive an online video clip, explaining the benefits of breastfeeding.
  Interventions: Behavioral: Video clip
- Control group (Sham Comparator): Participants will not receive the video clip
  Interventions: Behavioral: No video clip

INTERVENTIONS:
Behavioral: Video clip — After obtaining written informed consent, participants received a sealed envelope containing a preprinted paper referral to an online website, with a unique identifier.
  After entering the online website, participants will be asked to enter the unique identifier they have received into a text box. Only those whose identifiers were predetermined to be associated with the intervention group will receive the intervention.
  The intervention is twenty minutes long educational video clip, in which a brief discussion was presented, by an obstetrician, pediatrician, dietitian, and a breastfeeding consultant, each presenting the benefits of breastfeeding for mother and newborn.
  Other Names: Intervention group
  Arms: Educational video
Behavioral: No video clip — Participants in this group will receive a unique identifier that belongs to the control group, thus no video clip will be displayed.
  Other Names: Control group
  Arms: Control group

SUMMARY:
The goal of the study is to examine the impact of an educational video on the rate of breastfeeding in mothers who had gestational diabetes mellitus, and the rate of type-II diabetes mellitus diagnosed postpartum.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant individuals aged over 18 years old
* Diagnosed with Gestational Diabetes Mellitus (GDM) by 100gm oral glucose tolerance test (OGTT) done between week 24-28 of gestation, or by other criteria (50gm glucose challenge test (GCT) >200 mg/dl22 or having one abnormal value in OGTT )
* Having pregestational diabetes (DM-I or DM-II)
* Can read and understand Hebrew

Exclusion Criteria:

* Delivery of a non-viable fetus

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-05-30 (Estimated)

PRIMARY OUTCOMES:
Rate of type II Diabetes Mellitus (DM) diagnosis, as diagnosed by the 75gm oral glucose tolerance test (OGTT) | A phone call at 6 weeks postpartum.
  Participants are requested to perform 75gm oral glucose tolerance test (OGTT) postpartum, as a screening test for type I diabetes mellitus. We will record the results and compare between groups

SECONDARY OUTCOMES:
Rate of OGTT performance | A phone call at 6 weeks postpartum.
  Determination the actual performance of the test
Rate of impaired glucose tolerance (IGT) | A phone call at 6 weeks postpartum.
  Similar to primary outcome
Rate of exclusive breastfeeding | A phone call at 6 weeks postpartum.
  Participants will be asked by a phone cell, about feeding habits, including exclusive, partial and no breastfeeding of the infant

CONTACTS AND LOCATIONS:
Overall Officials: Nadav Cohen, MD, Principal Investigator — Carmel MC
Locations (1):
- Carmel MC, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gunderson EP, Hedderson MM, Chiang V, Crites Y, Walton D, Azevedo RA, Fox G, Elmasian C, Young S, Salvador N, Lum M, Quesenberry CP, Lo JC, Sternfeld B, Ferrara A, Selby JV. Lactation intensity and postpartum maternal glucose tolerance and insulin resistance in women with recent GDM: the SWIFT cohort. Diabetes Care. 2012 Jan;35(1):50-6. doi: 10.2337/dc11-1409. Epub 2011 Oct 19. PMID 22011407
- [Result] McFadden A, Gavine A, Renfrew MJ, Wade A, Buchanan P, Taylor JL, Veitch E, Rennie AM, Crowther SA, Neiman S, MacGillivray S. Support for healthy breastfeeding mothers with healthy term babies. Cochrane Database Syst Rev. 2017 Feb 28;2(2):CD001141. doi: 10.1002/14651858.CD001141.pub5. PMID 28244064